CLINICAL TRIAL: NCT00546403
Title: An Eight Week, Double-Blind, Placebo Controlled, Adjunctive Study of the Primary Effects of the Use of Flexible Doses of Modafinil 50mg to 200mg, on the Negative Symptoms, Cognition, and Excessive Daytime Sleepiness in Schizophrenic Patients
Brief Title: Modafinil Augmentation Therapy for Excessive Daytime Sleepiness and Negative Symptoms in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: Cephalon (Industry)
Responsible Party: James Lohr, MD, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1538a-633
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2007-10

CONDITIONS: Schizophrenia
Keywords: Excessive Daytime Sleepiness
MeSH Terms: conditions — Schizophrenia; Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Adjunctive treatment with placebo
  Interventions: Drug: Placebo
- Modafinil (Experimental): Treatment with titrated dose of study drug, modafinil.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Adjunctive treatment with titrated dose of modafinil
  Other Names: Provigil
  Arms: Modafinil
Drug: Placebo — Adjunctive treatment with placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effect of modafinil on the negative symptoms, such as blunted affect and social withdrawal, of schizophrenic patients and to determine modafinil's effect on excessive daytime sleepiness. A secondary purpose of the study is to examine the effect of modafinil on cognitive functioning of schizophrenic patients.

DETAILED DESCRIPTION:
Twenty six male patients with schizophrenia (twelve with Excessive Daytime Sleepiness and twelve without) will be enrolled at the San Diego Veterans Affairs Medical Center. Modafinil has been shown to increase alertness in individuals who are pathologically sleepy (Study C1538a/301/NAIUS).

Subjects will be randomized in a 1:1 ratio, stratified by excessive daytime sleepiness (value of >=9 on the Epworth Sleepiness Scale). Subjects will receive either modafinil or placebo, supplied by the sponsor. The study drug will be taken by mouth once daily in the morning. The titration schedule will be as follows:

1. The beginning does will be 50mg for 2 weeks
2. The study medication will be increased to 100mg at the week 2 study visit
3. The study medication will be increased to 200mg at the week 4 study visit and will continue for the remaining 4 weeks of the study. If subjects are unable to tolerate dosage increases, the dose will be decreased to the previous level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to communicate and give voluntary informed consent
* Subjects must be of the male gender
* Between the ages of 18 to 65 years.
* A diagnosis of Schizophrenia or Schizoaffective disorder as determined by DSM-IV criteria.
* Not conservatorized
* A negative symptom score on the PANSS of >= 20 and an MMSE score of >24
* No clinical evidence of a current unstable medical illness
* No current clinical evidence or past history of cerebral neurological impairment (including strokes, tumors or trauma leading to loss of consciousness)
* No history of drug or alcohol dependence in the past 2 years
* No evidence of drug or alcohol abuse in the past year, as determined by the DSM-IV criteria.
* No diagnosis of Narcolepsy as determined by DSM-IV criteria
* Must have an approved contact person for the duration of the study
* May be on a stable dose of SSRI for depressive symptoms
* No history of aggression
* No uncontrolled hypertension, as defined below (subjects cannot have any of the following):

  1. a new diagnosis of hypertension, or
  2. a change in antihypertensive medications in the past 30 days, or
  3. acute hypertension (systolic>160mmHg, diastolic>100mmHg)
* Maybe on a stable dose of a benzodiazepine
* The following medications will not be allowed during the study- methylphenidate, amphetamines, pemoline, zolpidem, MAO inhibitors, anticoagulant, TCA's, or barbiturates.
* Be on a stable does of an atypical neuroleptic
* May be on a stable does of an anticonvulsant for mood stabilization

Exclusion Criteria:

* Subjects cannot be female.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
PANSS, and Sleep/wake activity measured using the Actillume (Ambulatory Monitoring, Inc.) | baseline, one month, two months

SECONDARY OUTCOMES:
Neuropsychological Assessments that target cognitive abilities. | baseline, one month, two months

CONTACTS AND LOCATIONS:
Overall Officials: James B Lohr, MD, PhD, Principal Investigator — Director, VA Center of Excellence for Stress and Mental Health (CESAMH)
Locations (1):
- VA Healthcare System, Department of Psychiatry, San Diego, California, United States